CLINICAL TRIAL: NCT00463554
Title: An Evaluation of the GYNECARE TVT-SECUR* System (Tension-free Support for Incontinence) for the Treatment of Stress Urinary Incontinence *Trademark
Brief Title: TVT-SECUR A Pilot Study for the Treatment of Stress Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300-05-002
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Stress Urinary Incontinence
Keywords: Incontinence; Stress Urinary
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: GYNECARE TVT-SECUR* System — A sub-urethral sling for the treatment of SUI resulting from urethral hypermobility and/or intrinsic sphincter deficiency
  Other Names: Sub-urethral sling

SUMMARY:
The primary objective of this study is to obtain clinical performance information on the GYNECARE TVT-SECUR* System (Tension-free Support for Incontinence) in women with stress urinary incontinence (SUI).

DETAILED DESCRIPTION:
The primary variable for effectiveness is > 50% improvement on the subjective symptom Visual Analog Scale (VAS) at Visit 3/Week 5 (35 days post-surgery) to be accepted.

ELIGIBILITY:
Inclusion Criteria:

* Must be female with objective, demonstratable signs of SUI or stress predominant mixed incontinence and requires elective, primary surgical intervention.
* Must be at least 21 years old.
* Must be postmenopausal (amenorrhea) for at least 1 year or surgically sterile (bilateral salpingo-oophorectomy or tubal ligation or otherwise be incapable of pregnancy) or has a negative pregnancy test prior to study entry and has decided to cease childbearing.
* Agrees to participate in the study, including all study related procedures and evaluations and documents this agreement by signing the IRB/EC-approved informed consent

Exclusion Criteria:

* Have any other coexistent pathology requiring concomitant surgery that may impact this procedure i.e. surgeries that involve the anterior vaginal wall (e.g. anterior colporrhaphy, diverticula, anterior Prolift) Any allowable concomitant surgery must be performed prior to the GYNECARE TVT SECUR System surgery.
* Have intrinsic sphincter deficiency (ISD) [Urethral Pressure Profile (UPP) with a maximum urethral closing pressure (MUCP) < 20cm H2O or Leak Point Pressure (LPP) < 60].
* Have an active urinary tract infection (UTI) or vaginal infection at time of surgery.
* Have a fixed urethra (< 30° mobility on Q-Tip Straining Test).
* Have had prior incontinence surgery.
* Have a post-void residual volume > 100mL.
* Have co-existent pelvic organ prolapse that is symptomatic or extends beyond the hymen.
* Have lower urinary tract pathology in the form of a fistula or diverticulum.
* Have a malignancy or with a history of malignancy within the past 5 years, except for a basal cell carcinoma that has been treated with local excision and is no longer present.
* Are on anticoagulant therapy.
* Have received an experimental drug or used an experimental medical device within 30 days prior to the planned start of treatment.
* Are deemed by the investigator as medically unfit for surgery or who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications outlined in the GYNECARE TVT SECUR System IFU.
* Employees of the investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with stress urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance of TVT-SECUR* | Screening and Day 35

SECONDARY OUTCOMES:
Assessment of the results of the standing cough stress test | Screening, Week 5, Months 6 and 12
Intra- and post-operative complications | Intraoperative, Week 5, Months 6 and 12
Physician questionnaire results | Months 2 and 12
Urodynamics | Screening, Week 5, Months 6 and 12 (post-operative optional)
QoL measures | Screening, Week 5, Months 6 and 12
Subject satisfaction. | Month 12
Anesthesia | intraoperative
Operative time | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (6):
- United States (4):
  - Michigan Institute of Women's Health, Dearborn, Michigan
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Helsinki University Central Hospital, Helsinki, Finland
- University of Padova, Padua, Italy